CLINICAL TRIAL: NCT02095639
Title: Does Electroconvulsive Therapy Cause Neuroinflammation? An [18F]FEPPA Positron Emission Tomography Study in Treatment Resistant Depression
Brief Title: Inflammation and Electroconvulsive Therapy
Status: Terminated | Type: Observational
Why Stopped: The study was terminated
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Program Head, Neurochemical Imaging for Mood Disorders, Centre for Addiction and Mental Health
Other Study IDs: 074-2012
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma and serum samples will be kept for analysis of genotype, peripheral inflammatory markers and protein binding.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ECT and Treatment Resistant Depression: Subjects will be those with diagnosis of major depressive disorder that have not responded to many different treatments and who are planning to take electroconvulsive therapy (ECT). This group will receive two [18F]FEPPA PET scans, one baseline and one after an average of 2.5 weeks of ECT treatments.

SUMMARY:
The purpose of this study is to explore whether electroconvulsive therapy (ECT) accidentally leads to a side effect of brain inflammation. Patients with treatment resistant depression who are planning to take ECT will be subsequently approached to participate in the study.

DETAILED DESCRIPTION:
The first scan will take place before the first ECT session. The second scan will occur after a minimum of six ECT sessions (average 2.5 weeks). Secondary measures will include mood symptom severity, neurocognitive measures, peripheral inflammatory markers and TSPO genotype.

The hypothesis is that neuroinflammation will be increased by ECT.

There will be no alterations to standard care of depressed patients due to participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* stable physical health
* diagnosis of non-psychotic, non-catatonic, major depressive disorder, either unipolar or bipolar and a non-response to at least three clinical trials at appropriate dose of antidepressant medication from at least three different pharmacological classes
* at least a 17 on the17-item HDRS despite taking antidepressant treatment prior to ECT
* have not received ECT within the last 12 weeks

Exclusion Criteria:

* currently pregnant
* current substance abuse or dependence
* neurological or unstable medical illness
* use of anti-inflammatory drugs within the past month
* diazepam or other benzodiazepine use within the past month, except for lorazepam and clonazepam

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community and tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in translocator protein distribution volume (TSPO Vt) measured by [18F]FEPPA PET | Baseline scan and a second PET scan after an expected average time of 2.5 weeks of ECT treatment
  Participants will have one [18F]FEPPA PET scan before they start ECT and a second PET scan on average after 2.5 weeks of ECT

SECONDARY OUTCOMES:
17-item Hamilton Depression Rating Scale (HDRS) | Baseline and after average 2.5 weeks of ECT treatment
  Scores on the 17-item HDRS will be taken at the time of the PET scan (baseline and post-ECT) to assess whether the magnitude of change in TSPO distribution volume is associated with changes in symptom severity.
Neurocognitive Battery | Baseline and after average 2.5 to 5 weeks of ECT treatment
  Neurocognitive measures will be take at baseline and post-ECT to assess whether TSPO Vt is related to neurocognitive function. Neurocognitive battery includes:
  Autobiographical Memory Interview-Short Form (AMI-SF) Rey Auditory Verbal Learning Test (RAVLT) Wisconsin Card Sorting Test Comprehensive Trail Making Test Weschler Adult Intelligence Scale-Digit Symbol Subtest Stroop Color and Word Test Brief Visuospatial Memory Test Boston Naming Test Judgement of Line Orientation Weschler Test of Adult Reading
Peripheral Inflammatory Markers | Baseline and after average 2.5 to 5 weeks of ECT treatment
  To explore whether peripheral and central inflammation are related markers of peripheral inflammation (TNF-alpha, IL-6, CRP and IL-1beta) will be measured and correlated to brain TSPO Vt.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD, PhD, Principal Investigator — Research Imaging Centre, Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada